CLINICAL TRIAL: NCT05517564
Title: A Phase 1, First-in-Human, Double-blind, Placebo-controlled, Single-and Multiple-Ascending Oral Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of GM-60106 in Healthy Adults and Otherwise Healthy Adults With an Increased Body Mass Index and Markers of Non-Alcoholic Fatty Liver Disease
Brief Title: First-in-Human Study of GM-60106 in Healthy Adults and Otherwise Healthy Adults With an Increased Body Mass Index and Markers of Non-Alcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: JD Bioscience Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDB-106001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-08

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (GM-60106) (Experimental): Drug: GM-60106 Dosage: Part A: 2.5, 5, 10, 20, 40, 60, or 100 mg, Part B: 5, 10, 20 mg, Part C: 10, 20 mg Dosage Form: Bovine-gelatin capsules Route of Administration: Oral
  Interventions: Drug: GM-60106
- B (Placebo) (Experimental): Dosage Form: Bovine-gelatin capsules Route of Administration: Oral Matching placebo has an identical formulation to the GM-60106 drug product, prepared without the active pharmaceutical ingredient
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GM-60106 — The participants will receive a single oral dose between 2.5 to 100 mg for Part A (SAD), Part B (MAD) once daily for 14 days, and for Part C (MAD) once daily for 28 days.
  Arms: A (GM-60106)
Other: Placebo — Placebo-to-match GM-60106 capsules
  Arms: B (Placebo)

SUMMARY:
This is a Phase 1a/1b, randomised, double-blind, placebo-controlled single- and multiple-ascending dose study to evaluate the safety, tolerability, PK, and PD of GM-60106 in healthy adult male and female participants and otherwise healthy adults who have an increased BMI and markers of NAFLD.

DETAILED DESCRIPTION:
The study consists of 3 parts:

Part A (Single Ascending Dose [SAD]): Approximately 56 healthy participants will be enrolled into 7 cohorts and randomised to receive either GM-60106 or matching placebo at a ratio of 6:2 (GM-60106: placebo).

Part B (Multiple Ascending Dose [MAD]): Approximately 24 healthy participants will be enrolled into 3 cohorts and randomised to receive either GM-60106 or matching placebo at a ratio of 6:2 (GM-60106: placebo).

Part C (Multiple Ascending Dose [MAD]): Approximately 16 participants will be enrolled into 2 cohorts and randomised to receive either GM-60106 or matching placebo at a ratio of 6:2 (GM-60106: placebo). Cohorts will include otherwise healthy participants who have an increased BMI and markers of NAFLD.

Part B and Part C will occur only after the Safety Monitoring Committee (SMC) has reviewed all blinded safety data as well as any available PK and PD data from MAD cohorts that have completed the assessment of doses equal to the proposed starting Part C (MAD) dose and a dose higher (including a minimum safety review interval of 10 days after dosing the sixth participant in the cohort) and recommends initiation.

The study duration for each participant in Part A (SAD) is a maximum of 36 to 43 days, including a Screening period of up to 28 days, 1 day of single dosing, and a follow-up period of 7 days for most cohorts, and food effect assessment with a total treatment and follow-up period of 15 days for one of the SAD cohorts.

The study duration for each participant in Part B (MAD) is a maximum of 49 days, including a Screening period of up to 28 days, 14 consecutive days of once daily dosing, and a follow-up period of 7 days.

The study duration for each participant in Part C (MAD) is a maximum of 63 days, including a Screening period of up to 28 days, 28 consecutive days of once daily dosing, and a follow-up period of 7 days.

ELIGIBILITY:
Key inclusion Criteria:

1. Healthy adult males or females aged 18 to 55 years (inclusive)
2. Body weight ≥ 50 kg for males and ≥ 45 kg for females
3. Negative pregnancy test

Key exclusion criteria:

1. History or presence of clinically significant abnormalities or participants with psychosomatic disorders.
2. Positive test results for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) antibody.
3. Dosing in other clinical studies and treatment with a study drug within 3 months prior to IP administration.
4. Females who are pregnant or breastfeeding, or of childbearing potential who are not using effective non-hormonal contraception; men of childbearing potential who are unwilling to use physical methods of contraception during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess safety and tolerability of GM-60106 through incidence, nature, and severity of adverse events (AEs) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days

SECONDARY OUTCOMES:
The pharmacokinetics (PK) of GM-60106. Plasma sample will be collected for PK assessment. Parameter: maximum concentration (Cmax) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days
The pharmacokinetics (PK) of GM-60106. Plasma sample will be collected for PK assessment. Parameter: time to maximum concentration (Tmax) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days
The pharmacokinetics (PK) of GM-60106. Plasma sample will be collected for PK assessment. Parameter: Area under the curve (AUC) from time 0 to the last measurable concentration (AUC0-last) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days
The pharmacokinetics (PK) of GM-60106. Urine sample will be collected for PK assessment. Parameter: Cumulative amount of drug excreted in urine (Ae) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days
The pharmacokinetics (PK) of GM-60106. Urine sample will be collected for PK assessment. Parameter: Renal clearance (CLr). | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days
The pharmacodynamics (PD) of GM-60106 through liver function test (aspartate aminotransferase [AST]) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days
The pharmacodynamics (PD) of GM-60106 through liver function test (alanine aminotransferase [ALT]) | Part A: Up to 43 days, Part B: Up to 49 days, Part C: Up to 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Sam Francis, Principal Investigator — Nucleus Network Pty Ltd -Melbourne
Locations (2):
- Australia (2):
  - Nucleus Network Pty Ltd, Geelong, Victoria
  - Nucleus Network Pty Ltd, Melbourne, Victoria